CLINICAL TRIAL: NCT02051738
Title: A Single-Dose, Open-Label, Randomized, 2-Way Crossover Study to Assess the Effect of Food on the Bioavailability of Mebendazole From a Fast-Disintegrating Chewable Formulation of Mebendazole in Healthy Subjects
Brief Title: A Study to Assess the Effect of Food on the Bioavailability of Mebendazole From a Fast-Disintegrating Chewable Formulation of Mebendazole in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR103571; MEBENDAZOLGAI1002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2014-01-30; First posted 2014-01-31 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
Keywords: Healthy; Mebendazole; Fast-Disintegrating Chewable Formulation; Bioavailability
MeSH Terms: interventions — Mebendazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Sequence AB (Experimental): A single 500 mg dose of mebendazole fast-disintegrating chewable tablet will be administrated under fasted condition (Treatment A) in Treatment Period 1; In Treatment Period 2, the same medication will be administrated under fed condition (Treatment B).
  Interventions: Drug: Mebendazole - fasted state (Treatment A); Drug: Mebendazole - fed state (Treatment B)
- Treatment Sequence BA (Experimental): A single 500 mg dose of mebendazole fast-disintegrating chewable tablet will be administrated under fed condition (Treatment B) in Treatment Period 1; In Treatment Period 2, the same medication will be administrated under fasted condition (Treatment A).
  Interventions: Drug: Mebendazole - fasted state (Treatment A); Drug: Mebendazole - fed state (Treatment B)

INTERVENTIONS:
Drug: Mebendazole - fasted state (Treatment A) — Participants will receive a single 500 mg dose of mebendazole fast-disintegrating chewable tablet in the fasted condition.
  Other Names: VERMOX
Drug: Mebendazole - fed state (Treatment B) — Participants will receive a single 500 mg dose of mebendazole fast-disintegrating chewable tablet in the fed condition.
  Other Names: VERMOX

SUMMARY:
The purpose of the study is to evaluate the effect of food on the bioavailability (how much medication is in your blood) of mebendazole from a single 500 mg oral dose of a fast-disintegrating chewable tablet formulation of mebendazole in healthy adult participants.

DETAILED DESCRIPTION:
This is an open-label (the participant and the study physician know what the participant is getting), randomized (like the flip of a coin), single-center, single-dose, 2-way crossover (method used to switch participants from one treatment arm to another in a clinical study) study in approximately 16 healthy adult participants. Participants will receive study medication under fed state first and later under fasted state or vice versa. The study consists of 3 phases: screening phase of approximately 3 weeks, an open-label treatment phase consisting of two 6-day treatment periods (Treatment period 1 and 2) with a 7- to 10 day washout between Day 1 of each treatment period, and a safety follow-up phase occurring 7 to 10 days after the last study-related procedure on Day 5 of Treatment Period 2. The study physician will check participant's general health during the study. Total duration of study for each participant will be approximately 48 days.

ELIGIBILITY:
Inclusion Criteria:

* Must have signed an informed consent document
* Woman must be postmenopausal, surgically sterile, abstinent, or, if sexually active, be practicing an effective method of birth control before entry and throughout the study
* Woman must have a negative serum human chorionic gonadotropin pregnancy test at screening; and a negative urine pregnancy test on Day -1 of each treatment period
* Man must agree to use an adequate contraception method as deemed appropriate by the investigator and to not donate sperm during the study and for 3 months after receiving the last dose of study medication
* Blood pressure (after the participant is sitting for 5 minutes) between 90 and 140 mmHg systolic, inclusive, and no higher than 90 mmHg diastolic

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders, lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the subject or that could interfere with the interpretation of the study results
* Clinically significant abnormal values for hematology, clinical chemistry or urinalysis at screening or at admission to the study center on Day -1 of each Treatment Period as deemed appropriate by the investigator
* Clinically significant abnormal physical examination, vital signs or 12 lead electrocardiogram at screening or at admission to the study center on Day -1 of each Treatment Period as deemed appropriate by the investigator
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for paracetamol, oral contraceptives and hormonal replacement therapy within 14 days before dosing in each treatment period
* Positive test for drugs of abuse, such as cannabinoids, alcohol, opiates, cocaine, amphetamines, benzodiazepines, hallucinogens or barbiturates at screening and Day 1 of the each treatment period
* History of clinically significant allergies, especially known hypersensitivity or intolerance to lactose

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2014-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Concentration of mebendazole in blood and urine under fed and fasted condition | Up to Day 5 of in each treatment period

SECONDARY OUTCOMES:
Number of participants with adverse events | From screening up to 7 to 10 days after Day 5 of Treatment Period 2

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Merksem, Belgium